CLINICAL TRIAL: NCT00686400
Title: A German Multicenter Study on Toxoplasma Gondii in First-episode Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Silke Bachmann, MD, Dept. of Psychiatry, Psychotherapy and Psychosomatics, University of Halle
Other Study IDs: 07R-1815, SMRI
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder
Keywords: schizophrenia; first-episode; infection; Toxoplasma gondii; levels of IgG antibodies to TG
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, CSF if patients agree to lumbar puncture all frozen and stored at -80 degree Celsius until analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: FE: FE = first episode schizophrenia
  Interventions: Other: TAU = treatment as usual
- 2: CO: CO = age and gender-matched control subjects

INTERVENTIONS:
Other: TAU = treatment as usual — medication and psychosocial interventions to be chosen by treating psychiatrist
  Groups: 1: FE

SUMMARY:
Environmental risk factors for the development of schizophrenia include infections during the perinatal period or later in life with Toxoplasma gondii (TG) being one of the candidate agents. A recent review (Torrey and Yolken, 2003) on TG in schizophrenia and other serious mental disorder reported higher antibodies to TG in patients compared to controls in 18 of 19 studies, one having been conducted by the investigators group. In a second, independent study on first-episode schizophrenia (n=56) and control subjects (n=32), sera were sampled and standard instruments used to assess diagnoses and psychopathology, respectively to screening controls.

For the total sample, contacts with animals during pregnancy and age emerged as a non-significant predictors of TG IgG titers. Means of patients' and controls' TG IgG titers did not differ significantly but variances did; a subgroup of patients' titers reached much higher levels than those of controls. Patients in the high TG IgG subgroup were older (p=0.001), also they were older when psychiatric symptoms appeared, more individuals had regular animal contacts during pregnancy, or rural upbringing including regular animal contact, more consumption of raw meat, and a higher absolute treatment response (all trend levels). Regarding the short term course of patients, the investigators detected decreasing IgG titers in several individuals A power analysis demonstrated that results fell short of significance due to lack of statistical power. Based on the power analysis, the investigators propose an opel label, multicenter study at three regionally different sites within Germany (Halle, Hamm, Heidelberg). The investigators intent to study 173 first-episode patients with schizophrenia, schizoaffective, and schizophreniform disorder and 173 matched controls.

The investigators hypothesize that - according to the heterogeneity of the illness - a subgroup of patients will exhibit higher TG IgG titers compared to the remaining patients and to controls; that this subgroup will have had regular contact with animals during pregnancy and early life as well as developmental delays; and that clinical improvement, response to treatment, and subjective well-being will run parallel with TG IgG decrease.

Patients shall be assessed on admission to hospital, at discharge and at 6- and 12-month-follow-up with respect to TG antibody titers, symptomatology, neuropsychology, predictors of outcome, quality of life, and neurological soft signs. In controls two assessments shall be performed, 12 months apart. All foreseen assessments will be performed using standard measurement instruments with sound reliability and validity such as the SCID and the PANSS. Exposure to cats, other warm-blooded life-stock, and raw meat will be assessed using a special questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria will be a first episode of schizophrenia, schizoaffective or schizophreniform disorder.

Exclusion Criteria:

* Exclusion criteria will be major organic and substance induced disorders, refusal or withdrawal of IC.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who are admitted to inpatient treatment due to a first episode of psychotic symptoms, diagnoses of schizophrenia, schizophreniform and schizoaffective disorder age- and gender-matched control subjects
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-12 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
falling levels of Toxoplasma IgG titers parallel clinical improvement over time, 2 follow-ups at 6 and 12 months are planned | 3 years

SECONDARY OUTCOMES:
clinical improvement; outcome: functioning and psychopathology | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Silke Bachmann, MD, assistant prof. psychiatry, Principal Investigator — Dept. of Psychiatry, Psychotherapy and Psychosomatics, University of Halle (Saale), Germany
Locations (3):
- Germany (3):
  - Dpt. of Psychiatry, University of Frankfurt, Frankfurt am Main
  - Dept. of Psychiatry, University of Halle (Saale), Halle
  - Dept. of Psychiatry, University of Heidelberg, Heidelberg

REFERENCES:
- [Background] Torrey EF, Yolken RH. Toxoplasma gondii and schizophrenia. Emerg Infect Dis. 2003 Nov;9(11):1375-80. doi: 10.3201/eid0911.030143. PMID 14725265
- [Background] Yolken RH, Bachmann S, Ruslanova I, Lillehoj E, Ford G, Torrey EF, Schroeder J. Antibodies to Toxoplasma gondii in individuals with first-episode schizophrenia. Clin Infect Dis. 2001 Mar 1;32(5):842-4. doi: 10.1086/319221. Epub 2001 Feb 28. PMID 11229859
- [Background] Bachmann S, Schroder J, Bottmer C, Torrey EF, Yolken RH. Psychopathology in first-episode schizophrenia and antibodies to Toxoplasma gondii. Psychopathology. 2005 Mar-Apr;38(2):87-90. doi: 10.1159/000085349. Epub 2005 Apr 22. PMID 15855832
- See also: The SMRI funds this study, sample analyses wil be made at the Stanley Laboratory of Developmental Neurovirology at the Johns Hopkins University, Baltimore, MD, USA — http://www.stanleyresearch.org